CLINICAL TRIAL: NCT00956254
Title: Evaluate Safety and Tolerability and Compare Absorption/Distribution Kinetics of a Single 100 Mcg Dose of Fentanyl Sublingual Spray (Fentanyl SL Spray) in Cancer Subjects With or Without Oral Mucositis
Brief Title: Fentanyl Sublingual Spray in Treating Opioid-tolerant Cancer Patients With or Without Oral Mucositis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INS-09-011; CDR0000647007 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-06

CONDITIONS: Mucositis; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: mucositis; unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Mucositis; Pain

ARMS (1):
- Fentanyl sublingual spray 100 µg (Experimental): Participants received a single administration of fentanyl sublingual spray 100 µg sublingually.
  Interventions: Drug: Fentanyl sublingual spray

INTERVENTIONS:
Drug: Fentanyl sublingual spray — Fentanyl was supplied in single-dose glass vials assembled into a delivery device to be used as a sublingual spray.

SUMMARY:
This was an open-label, single-dose study to assess the safety, tolerability, and absorption/distribution kinetics of a single 100 µg dose of fentanyl sublingual spray in opioid-tolerant cancer subjects, with or without oral mucositis.

DETAILED DESCRIPTION:
RATIONALE: One dose of fentanyl sublingual spray may be effective in relieving pain in opioid-tolerant cancer patients.

PURPOSE: This phase III trial is studying the side effects of fentanyl sublingual spray and to see how well it works in treating opioid-tolerant cancer patients with or without oral mucositis.

OBJECTIVES:

Primary

* To compare the absorption/distribution kinetics of a single dose of fentanyl sublingual spray in opioid-tolerant cancer patients with or without oral mucositis.
* To evaluate the safety and tolerability of this regimen.

OUTLINE: This is a multicenter study.

Patients fast for at least 8 hours before and at least 4 hours after and no water is allowed for at least 1 hour before and at least 1 hour after study drug administration. Patients receive a single dose of fentanyl sublingual spray while in an upright position in clinical care recliners or beds, and remain in an upright posture for at least 4 hours after administration. Patients are instructed not to swallow for at least 5 minutes after administration and not to expectorate the drug.

After study drug administration, 10 blood samples are collected over a 12-hour period for pharmacokinetic and other analyses.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer and meets 1 of the following criteria:

  * Mild mucositis, defined as grade 1 (erythema of the mucosa) or 2 (patchy ulcerations or pseudomembranes) on the day of study drug administration.
  * No mucositis, defined as normal oral cavity upon examination on the day of study drug administration.
* Opioid-tolerant, defined as patients who are taking ≥ 60 mg of oral morphine/day, ≥ 30 mg of oxycodone/day, ≥ 8 mg of oral hydromorphone/day, or an equianalgesic dose of another opioid for ≥ 7 days for cancer-related pain.
* Persistent pain related to cancer or its treatment over the past 7 days.
* No brain metastases with signs or symptoms of increased intracranial pressure.

PATIENT CHARACTERISTICS:

* Negative pregnancy test.
* Agree to be confined to study site for approximately 12 hours, to eat only the food served by the study unit during the study confinement period, and to consume all food provided at the designated meal or snack times.
* No history of major organ system impairment or disease that, in the investigator's or his/her designee's opinion, could increase the risk associated with the use of opioids.
* No uncontrolled hypertension despite antihypertensive therapy or history of hypertensive crisis within the past 2 years.
* No recent history (within the past 2 years) of transient ischemic attacks, neural vascular disease, stroke, or cerebral aneurysms.
* No intolerable side effects to opioids or fentanyl.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics.
* More than 30 days since prior investigational agents.
* More than 14 days since prior monoamine oxidase inhibitors.
* No prior participation in either Insys Fentanyl Sublingual Spray Phase III study INSYS-INS-05-001 or INSYS-INS-06-007.
* No other concurrent use of any fentanyl product.

  * Patients who have received Actiq®, Fentora®, or Duragesic® are eligible after a 7-day washout.
* No concurrent medications (prescription, over-the-counter, vitamin, or herbal substances) except for hormonal contraceptives and/or ≤ 3 doses of acetaminophen at ≤ 1 g each.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J. Stearns, MD, Principal Investigator — Center for Pain and Supportive Care, PLLC
Locations (1):
- InSys Therapeutics, Incorporated, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fentanyl Sublingual Spray 100 µg
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All subjects who received study drug.
Arm/Group | Fentanyl Sublingual Spray 100 µg
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Fentanyl
Description: Cmax is defined as the maximum drug concentration in plasma and was determined from individual plasma concentration versus time data. Blood samples for pharmacokinetic analysis were drawn pre-dose; 15 and 30 minutes; and 1, 2, 4, 6, 8, 10, and 12 hours post-dose. Fentanyl concentration assays were performed using a fully validated and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Results are reported for patients with and without mucositis.
Time Frame: Pre-dose to 12 hours post-dose
Population: Pharmacokinetic (PK) population: All subjects who had evaluable plasma profiles to calculate reliable estimates of PK parameters and who had no major protocol deviations. One subject in the non-mucositis group self-administered a fentanyl product before receiving the study drug and was excluded from the PK population due to this protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fentanyl Sublingual Spray 100 µg - Mucositis; Fentanyl Sublingual Spray 100 µg - Non-mucositis: Participants received a single administration of fentanyl sublingual spray 100 µg sublingually.
Arm/Group | Fentanyl Sublingual Spray 100 µg - Mucositis | Fentanyl Sublingual Spray 100 µg - Non-mucositis
Number analyzed (Participants) | 9 | 8
ng/mL | 0.67 (0.60) | 0.26 (0.15)

2. Secondary Outcome: Tmax of Fentanyl
Description: Tmax is defined as the time to reach the maximum concentration of fentanyl in plasma and was determined from individual concentration versus time data. Blood samples for pharmacokinetic analysis were drawn pre-dose; and 15 and 30 minutes; and 1, 2, 4, 6, 8, 10, and 12 hours post-dose. Fentanyl concentration assays were performed using a fully validated and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Results are reported for patients with and without mucositis.
Time Frame: Pre-dose to 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Fentanyl Sublingual Spray 100 µg - Mucositis | Fentanyl Sublingual Spray 100 µg - Non-mucositis
Number analyzed (Participants) | 9 | 8
hr | 0.53 (0.57) | 0.56 (0.59)

3. Secondary Outcome: AUC0-last of Fentanyl
Description: AUC0-last is defined as the area under the plasma concentration-time curve from time-zero to the time of the last quantifiable concentration of fentanyl, was calculated using the linear trapezoidal rule, and was determined from individual concentration versus time data. Blood samples for pharmacokinetic analysis were drawn pre-dose; and 15 and 30 minutes; and 1, 2, 4, 6, 8, 10, and 12 hours post-dose. Fentanyl concentration assays were performed using a fully validated and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Results are reported for patients with and without mucositis.
Time Frame: Pre-dose to 12 hours post-dose
Population: Pharmacokinetic evaluable population: All subjects who had evaluable plasma profiles to calculate reliable estimates of pharmacokinetic parameters and who had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Fentanyl Sublingual Spray 100 µg - Mucositis | Fentanyl Sublingual Spray 100 µg - Non-mucositis
Number analyzed (Participants) | 9 | 8
hr*ng/mL | 3.11 (4.80) | 0.91 (0.13)

ADVERSE EVENTS:
Description: Safety population: All subjects who received study drug.
Arm/Group | Fentanyl Sublingual Spray 100 µg - Mucositis | Fentanyl Sublingual Spray 100 µg - Non-mucositis
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Sublingual Spray 100 µg - Mucositis (N=9) | Fentanyl Sublingual Spray 100 µg - Non-mucositis (N=9)
Burning sensation mucosal (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No